CLINICAL TRIAL: NCT06368349
Title: Persistent Lymphopenia as a Prognostic Indicator in Liver Transplantation and Its Molecular Insights for Hepatocellular Carcinoma Recipients
Brief Title: Persistent Lymphopenia in Liver Transplantation and Its Molecular Insights for Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202101771B0
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2021-10

CONDITIONS: Lymphopenia
Keywords: Liver transplantation; immune cell subtype; immunosuppressant
MeSH Terms: conditions — Lymphopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A total of 145 Liver transplantation (LT) recipients with hepatocellular carcinoma (HCC) were retrospectively enrolled at Kaohsiung Chang Gung Memorial Hospital between 2006 and 2019. Clinical records from 7 days before LT (pre-LT) to 1 year after LT (post-LT) were analysed. In a prospective study from March 2022 to June 2023, 20 lymphopenia and 25 non-lymphopenia HCC recipients were enrolled, and a phenotypic analysis of peripheral blood lymphocytes was performed using multiparameter flow cytometry.

DETAILED DESCRIPTION:
A total of 145 Liver transplantation (LT) recipients with hepatocellular carcinoma (HCC) were retrospectively enrolled at Kaohsiung Chang Gung Memorial Hospital between 2006 and 2019. Clinical records from 7 days before LT (pre-LT) to 1 year after LT (post-LT) were analysed including overall survival, recurrence-free survival, association between clinical parameter with mortality, patient characteristics by pre-lymphopenia and post-lymphopenia levels and lymphocyte status of HCC patients with usage of different immunosuppressants. In prospective study from March 2022 to June 2023, 20 lymphopenia and 25 non-lymphopenia HCC recipients were enrolled, and a phenotypic analysis of peripheral blood lymphocytes was performed using multiparameter flow cytometry to identify the major immune cell subsets and the characteristics of patients in the prospective cohort between pre-LT lymphopenia and non-lymphopenia groups.

ELIGIBILITY:
Inclusion Criteria:

* liver transplant patient

Exclusion Criteria:

* End-stage liver disease scoring system score (MELD score) > 25
* Have received care in the intensive care unit (ICU) before transplantation
* Poor cardiovascular function.
* Patients suffering active infection.
* Other complications affecting living donor liver transplantation

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 190 Liver transplantation (LT) recipients were enrolled including 145 cases for retrospective and 45 cases for perspective
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Persistent lymphopenia predict poor overall survival | From 2006 to 2019
  The clinical records of 145 patients with HCC from seven days pre-LT to one-year post-LT illustrated that the longitudinal values of lymphocytes were persistently low in patients with peritransplant high neutrophil lymphocyte ratio, indicating a significant decrease in survival rate when compared to other patients.
T cell and its subtype were mainly decrease in pre-LT lymphopenia population of HCC patient | From March 2022 to June 2023
  A significant decrease in cell counts and percentage of overall T cells in the peritransplant lymphopenia group. In particular, the counts of T cell subsets, T helper cells, and cluster of differentiation 8 (CD8+) cytotoxic/activated T cells significantly decreased in the peritransplant lymphopenia group with all of their naïve, effector, and memory forms.
Long-term peri-LT lymphopenia HCC recipients is associated with increased sirolimus use and decreased tacrolimus use | From 2006 to 2019
  In the subset of 116 of 145 HCC recipients (80%) who did not experience or recover from lymphopenia, no significant associations were observed with immunosuppressant use. Surprisingly, HCC recipients with long-term peritransplant lymphopenia exhibited a significant association with increased sirolimus use (p = 0.024) and decreased tacrolimus use (p = 0.001), whereas those with post-LT lymphopenia showed no association with the use of different immunosuppressants.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Kaohsiung City, Taiwan

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT06368349/Prot_SAP_000.pdf